CLINICAL TRIAL: NCT04363645
Title: Case Studies: Promoting Strategy Use in Functional Activities
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: New York Presbyterian Hospital (Other); Mercy University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1308014257
Record Dates: First submitted 2020-04-23; First posted 2020-04-27 (Actual); Last update posted 2020-04-27 (Actual); Status verified 2020-04

CONDITIONS: Cognitive Impairment; Executive Dysfunction; Acquired Brain Injury
MeSH Terms: conditions — Cognitive Dysfunction; Brain Injuries

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Multicontext approach (Intervention) Arm (Experimental): Participants received 30-minute sessions of strategy and self-monitoring practice within the context of everyday activities. These sessions were delivered either daily or twice a day. The total number of sessions varied depending on the participant's length of stay in acute rehabilitation.
  Interventions: Other: Multicontext (MC) approach

INTERVENTIONS:
Other: Multicontext (MC) approach — The Multicontext approach is a metacognitive intervention designed to improve awareness, strategy use, and executive functioning.

SUMMARY:
The purpose of the study is to provide evidence of feasibility, acceptability, patient satisfaction, and patient perceived benefit of the Multicontext (MC) approach. The project consists of eight case studies of persons with acquired brain injury undergoing acute inpatient rehabilitation who have difficulties in completing multiple step activities due to deficits in executive function and/or visual perception. The MC approach provides a structured occupational therapy framework that provides guidelines for enhancing strategy use and self monitoring skills for person's with acquired brain injury.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 80 years
* English-speaking
* Confirmed diagnosis of acquired brain injury (ABI) based on radiological assessment
* Able to comprehend multistep directions and participate in conversation as assessed by the Functional Independence Measure (FIM; required score of 4 or above on Comprehension and Expression items)
* Impaired performance (<2 SD below demographically-corrected normative data) on at least one screening measure of executive functioning
* Able to attend to a cognitive task for at least 10 minutes
* Cognitively independent in basic self-care activities
* Able to read standard size newsprint
* Ability to demonstrate functional use of at least one hand.

Exclusion Criteria:

* Global aphasia or moderate - severe comprehension deficits (as indicated by a FIM comprehension score of less than 4)
* Global cognitive impairment or dementia as indicated by a score of 20 or less on the Montreal cognitive assessment
* History of treatment for substance abuse or hospitalizations for psychiatric disorder, within the past year
* non-English speaking

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2014-12-14 (Actual); Primary Completion 2016-12-29 (Actual); Study Completion 2016-12-29 (Actual)

PRIMARY OUTCOMES:
Patient satisfaction, as measured by the Patient Satisfaction Questionnaire | End of study (approximately 2 weeks)
  The Patient Satisfaction Questionnaire consists of open-ended questions of what participants liked most and least about the program, what they would have changed about the program, and any additional suggestions or recommendations. This questionnaire also included Likert-type ratings of their satisfaction, enjoyment, perceived benefit from the intervention, and perceived likelihood of continuing to use the strategies learned in treatment. Patient satisfaction is qualitatively evaluated.
Change from baseline in metacognitive skills, as measured by the Self-Regulation Skills Interview (SRSI) | Baseline, end of study (approximately 2 weeks)
  The SRSI is a clinician-administered semi-structured interview that assesses an individual's metacognitive skills and ability to use cognitive strategies. It comprises six questions and each question is scored on a 10-point Likert-type scale. It consists of a total score and three factors, Awareness, Readiness to Change, and Strategy Behavior. The total score ranges from 0 to 60, with lower scores indicating greater metacognitive skills.
Change from baseline in executive functioning, as measured by the Weekly Calendar Planning Activity (WCPA) | Baseline, end of study (approximately 2 weeks)
  The WCPA is a standardized, performance-based, ecologically-valid measure of executive functioning in which the participant has to organize a list of appointments into a weekly schedule. The outcome variable is the percentage of appointments entered correctly relative to the total number of appointments entered.
Change from baseline in disability, as measured by the Functional Independence Measure (FIM) | Baseline, end of study (approximately 2 weeks)
  The FIM is a standard-of-care measure of disability that assesses the level of assistance required for an individual to perform activities of daily living. The FIM is comprised of 18 items. Each item is rated on a 1-7 scale. The FIM Total scores range from 18 to 126, with higher scores indicating greater functional independence.

CONTACTS AND LOCATIONS:
Overall Officials: Michael W O'Dell, M.D., Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medicine, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Jaywant A, Steinberg C, Lee A, Toglia J. Feasibility and acceptability of the multicontext approach for individuals with acquired brain injury in acute inpatient rehabilitation: A single case series. Neuropsychol Rehabil. 2022 Mar;32(2):211-230. doi: 10.1080/09602011.2020.1810710. Epub 2020 Sep 2. PMID 32873157